CLINICAL TRIAL: NCT07406685
Title: The Comparison of Ibandronate and Zoledronic Acid After Denosumab Discontinuation: A Randomized Non-inferiority Trial
Brief Title: The Comparison of Ibandronate and Zoledronic Acid After Denosumab Discontinuation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202601190MINA
Record Dates: First submitted 2026-02-01; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Postmenopausal Osteoporosis; Postmenopausal Osteopenia; Primary Osteoporosis; Osteoporosis
Keywords: Postmenopausal; Osteoporosis; Osteopenia; Denosumab; Ibandronate; Zoledronic acid; Discontinuation
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibandronate group (Experimental): use Ibandronate 1 year and follow-up for 2 years
  Interventions: Drug: Ibandronate IV
- Zoledronic acid group (Active Comparator): use Zoledronic acid 1 year and follow-up for 2 years
  Interventions: Drug: Zoledronic acid IV

INTERVENTIONS:
Drug: Ibandronate IV — Ibandronate 3mg/3months for 12 months
  Arms: Ibandronate group
Drug: Zoledronic acid IV — Zoledronic acid 5mg/1year for 12 months
  Arms: Zoledronic acid group

SUMMARY:
This study is a prospective, multicenter, open-label, randomized non-inferiority trial comparing intravenous ibandronate and zoledronic acid as sequential therapy after denosumab discontinuation in postmenopausal women with osteoporosis. This trial primarily targets patients with short-term denosumab exposure (less than three years) and is conducted as a preliminary investigation. The findings are expected to provide foundational evidence to inform the design of future studies assessing sequential therapies following longer-term denosumab treatment.

DETAILED DESCRIPTION:
Osteoporosis has been recognized by the World Health Organization (WHO) as the second most prevalent global epidemic disease, following coronary heart disease. Untreated osteoporosis may lead to a vicious cycle of recurrent fractures, resulting in disability and even mortality. In clinical practice, antiresorptive agents are commonly used as first-line therapy. Denosumab is widely preferred due to its convenient administration and potent suppression of bone turnover. However, its antiresorptive effect is reversible; discontinuation of denosumab is associated with rebound increases in bone turnover markers (BTMs) and rapid bone mineral density (BMD) loss. Therefore, subsequent antiresorptive therapy is required to prevent fracture occurrence. Zoledronic acid has been shown to effectively suppress post-denosumab rebound bone turnover and is currently considered the standard sequential treatment following denosumab discontinuation.

The objective of this study is to demonstrate that ibandronate, when used as a sequential therapy after denosumab discontinuation, provides protection comparable to zoledronic acid in patients with short-term denosumab exposure (< 3 years). This study aims to generate preliminary clinical evidence to support future trials and to offer an alternative post-denosumab treatment strategy in clinical practice. Participants will receive one year of ibandronate or zoledronic acid therapy, initiated 6 months (± 1 week) after the last dose of denosumab, followed by a total of two years of follow-up. Eligible participants will be randomized in a 1:1 ratio, with an estimated sample size of 26 patients per group.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women aged 50 to 85 years.
2. BMD T-score ≤ -1.5 and > -3.0 at the lumbar spine or total hip.
3. Regular treatment with denosumab administered every 6 months for at least 1 year and less than 3 years (3 to 5 doses).
4. Physically and mentally capable of understanding and complying with the study protocol and follow-up.
5. Signed informed consent.

Exclusion Criteria:

1. History of fragility or osteoporotic fracture within the past 12 months.
2. Current or prior treatment within the past 12 months with osteoporosis medications other than denosumab, including Romosozumab, Teriparatide, Alendronate, Ibandronate, Zoledronic acid, Risedronate and Raloxifene.
3. Allergy to bisphosphonates.
4. Secondary osteoporosis.
5. Metabolic bone diseases.
6. Any autoimmune disease.
7. Requirement for long-term use of medications known to affect bone metabolism (e.g., systemic glucocorticoids or hormone therapy).
8. Primary or metastatic bone tumors.
9. Cancer patients, except for in situ carcinoma and non-melanoma skin cancer, unless fully treated and in remission for five years.
10. Hypocalcemia.
11. Vitamin D deficiency (serum 25-hydroxyvitamin D < 25 ng/mL).
12. Renal disease (eGFR < 35 mL/min/1.73 m²) or dialysis patients.
13. Planned dental procedures (e.g., extractions, implants) within the next year.
14. Smoking more than one pack per day (except for those who have quit for over ten years).

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-03-17 (Estimated); Primary Completion 2030-03-17 (Estimated); Study Completion 2030-09-17 (Estimated)

PRIMARY OUTCOMES:
Percentage change in bone mineral density (BMD) | Baseline to 24 months after treatment initiation.
  Change in BMD at the lumbar spine, femoral neck, and total hip measured by dual-energy X-ray absorptiometry (DXA) from baseline to 24 months.
  Baseline is defined as the time point 6 months after the last dose of denosumab, immediately prior to initiation of sequential therapy. BMD measurements will be performed at 6, 12, 18, and 24 months after treatment initiation.

SECONDARY OUTCOMES:
Change in bone turnover makers (BTM) level | Baseline to 24 months
  Changes in serum bone turnover markers, including procollagen type 1 N-terminal propeptide (P1NP) and C-terminal telopeptide of type I collagen (CTX), will be evaluated to assess bone metabolic activity following denosumab discontinuation and sequential therapy.
  Measurements will be obtained at baseline and at 3, 6, 9, 12, 18, and 24 months after treatment initiation.
Change in visual Analogue Scale (VAS) score | Baseline to 24 months
  The Visual Analogue Scale (VAS) for pain will be used to assess participants' self-reported pain intensity. The VAS score ranges from 0 to 10, higher scores indicate worse pain intensity, and lower scores indicate less pain.
  Pain intensity of the lower back and lower extremities will be evaluated at baseline and every 6 months during follow-up.
Incidence of osteoporotic fractures | During the intervention period, up to 24 months.
  The occurrence and anatomical sites of osteoporotic fractures will be recorded throughout the study period.
Incidence of adverse events (AEs) and serious adverse events (SAEs) | During the intervention period, up to 24 months.
  All AEs and SAEs will be recorded and evaluated throughout the study period to assess the safety of sequential therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kumar S, Wang M, Kim AS, Center JR, McDonald MM, Girgis CM. Denosumab discontinuation in the clinic: implications of rebound bone turnover and emerging strategies to prevent bone loss and fractures. J Bone Miner Res. 2025 Aug 24;40(9):1017-1034. doi: 10.1093/jbmr/zjaf037. PMID 40057981
- [Result] Ha J, Jung KY, Kim KJ, Ahn SH, Kim HJ, Chung YS. Effects of Sequential Anti-Resorptive Agents on Bone Mineral Density Following Denosumab Withdrawal: A Multicenter Real-World Study in Korea (MAXCARE Study). Endocrinol Metab (Seoul). 2025 Oct;40(5):748-758. doi: 10.3803/EnM.2024.2227. Epub 2025 Feb 11. PMID 39933434
- [Result] Ramchand SK, Tsai JN, Lee H, Sassana-Khadka G, Jordan M, Ryan S, Leder BZ. The comparison of alendronate and raloxifene after denosumab (CARD) study: A comparative efficacy trial. Osteoporos Int. 2024 Feb;35(2):255-263. doi: 10.1007/s00198-023-06932-2. Epub 2023 Oct 6. PMID 37798320
- [Result] Kendler D, Chines A, Clark P, Ebeling PR, McClung M, Rhee Y, Huang S, Stad RK. Bone Mineral Density After Transitioning From Denosumab to Alendronate. J Clin Endocrinol Metab. 2020 Mar 1;105(3):e255-64. doi: 10.1210/clinem/dgz095. PMID 31665314
- [Result] Lee CC, Wang CY, Yen HK, Hung CC, Lai CY, Hu MH, Wang TM, Li CY, Fu SH. Zoledronate Sequential Therapy After Denosumab Discontinuation to Prevent Bone Mineral Density Reduction: A Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2443899. doi: 10.1001/jamanetworkopen.2024.43899. PMID 39527056
- [Result] Tutaworn T, Nieves JW, Wang Z, Levin JE, Yoo JE, Lane JM. Bone loss after denosumab discontinuation is prevented by alendronate and zoledronic acid but not risedronate: a retrospective study. Osteoporos Int. 2023 Mar;34(3):573-584. doi: 10.1007/s00198-022-06648-9. Epub 2023 Jan 5. PMID 36602607
- [Result] Solling AS, Harslof T, Langdahl B. Treatment With Zoledronate Subsequent to Denosumab in Osteoporosis: A 2-Year Randomized Study. J Bone Miner Res. 2021 Jul;36(7):1245-1254. doi: 10.1002/jbmr.4305. Epub 2021 Apr 20. PMID 33813753
- [Result] Anastasilakis AD, Papapoulos SE, Polyzos SA, Appelman-Dijkstra NM, Makras P. Zoledronate for the Prevention of Bone Loss in Women Discontinuing Denosumab Treatment. A Prospective 2-Year Clinical Trial. J Bone Miner Res. 2019 Dec;34(12):2220-2228. doi: 10.1002/jbmr.3853. Epub 2019 Oct 14. PMID 31433518
- [Result] Burckhardt P, Faouzi M, Buclin T, Lamy O; The Swiss Denosumab Study Group. Fractures After Denosumab Discontinuation: A Retrospective Study of 797 Cases. J Bone Miner Res. 2021 Sep;36(9):1717-1728. doi: 10.1002/jbmr.4335. Epub 2021 May 19. PMID 34009703
- [Result] Cosman F, Huang S, McDermott M, Cummings SR. Multiple Vertebral Fractures After Denosumab Discontinuation: FREEDOM and FREEDOM Extension Trials Additional Post Hoc Analyses. J Bone Miner Res. 2022 Nov;37(11):2112-2120. doi: 10.1002/jbmr.4705. Epub 2022 Oct 12. PMID 36088628
- [Result] Cummings SR, Ferrari S, Eastell R, Gilchrist N, Jensen JB, McClung M, Roux C, Torring O, Valter I, Wang AT, Brown JP. Vertebral Fractures After Discontinuation of Denosumab: A Post Hoc Analysis of the Randomized Placebo-Controlled FREEDOM Trial and Its Extension. J Bone Miner Res. 2018 Feb;33(2):190-198. doi: 10.1002/jbmr.3337. Epub 2017 Nov 22. PMID 29105841
- [Result] Anastasilakis AD, Polyzos SA, Makras P, Aubry-Rozier B, Kaouri S, Lamy O. Clinical Features of 24 Patients With Rebound-Associated Vertebral Fractures After Denosumab Discontinuation: Systematic Review and Additional Cases. J Bone Miner Res. 2017 Jun;32(6):1291-1296. doi: 10.1002/jbmr.3110. Epub 2017 Mar 13. PMID 28240371
- [Result] Bone HG, Wagman RB, Brandi ML, Brown JP, Chapurlat R, Cummings SR, Czerwinski E, Fahrleitner-Pammer A, Kendler DL, Lippuner K, Reginster JY, Roux C, Malouf J, Bradley MN, Daizadeh NS, Wang A, Dakin P, Pannacciulli N, Dempster DW, Papapoulos S. 10 years of denosumab treatment in postmenopausal women with osteoporosis: results from the phase 3 randomised FREEDOM trial and open-label extension. Lancet Diabetes Endocrinol. 2017 Jul;5(7):513-523. doi: 10.1016/S2213-8587(17)30138-9. Epub 2017 May 22. PMID 28546097
- [Result] Bone HG, Bolognese MA, Yuen CK, Kendler DL, Miller PD, Yang YC, Grazette L, San Martin J, Gallagher JC. Effects of denosumab treatment and discontinuation on bone mineral density and bone turnover markers in postmenopausal women with low bone mass. J Clin Endocrinol Metab. 2011 Apr;96(4):972-80. doi: 10.1210/jc.2010-1502. Epub 2011 Feb 2. PMID 21289258
- [Result] Cummings SR, San Martin J, McClung MR, Siris ES, Eastell R, Reid IR, Delmas P, Zoog HB, Austin M, Wang A, Kutilek S, Adami S, Zanchetta J, Libanati C, Siddhanti S, Christiansen C; FREEDOM Trial. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med. 2009 Aug 20;361(8):756-65. doi: 10.1056/NEJMoa0809493. Epub 2009 Aug 11. PMID 19671655
- [Result] Miller PD, Bolognese MA, Lewiecki EM, McClung MR, Ding B, Austin M, Liu Y, San Martin J. Effect of denosumab on bone density and turnover in postmenopausal women with low bone mass after long-term continued, discontinued, and restarting of therapy: a randomized blinded phase 2 clinical trial. Bone. 2008 Aug;43(2):222-229. doi: 10.1016/j.bone.2008.04.007. Epub 2008 Apr 26. PMID 18539106
- [Result] Black DM, Bauer DC, Vittinghoff E, Lui LY, Grauer A, Marin F, Khosla S, de Papp A, Mitlak B, Cauley JA, McCulloch CE, Eastell R, Bouxsein ML; Foundation for the National Institutes of Health Bone Quality Project. Treatment-related changes in bone mineral density as a surrogate biomarker for fracture risk reduction: meta-regression analyses of individual patient data from multiple randomised controlled trials. Lancet Diabetes Endocrinol. 2020 Aug;8(8):672-682. doi: 10.1016/S2213-8587(20)30159-5. PMID 32707115
- [Result] Fogelman I, Blake GM. Different approaches to bone densitometry. J Nucl Med. 2000 Dec;41(12):2015-25. PMID 11138687
- [Result] LeBoff MS, Greenspan SL, Insogna KL, Lewiecki EM, Saag KG, Singer AJ, Siris ES. The clinician's guide to prevention and treatment of osteoporosis. Osteoporos Int. 2022 Oct;33(10):2049-2102. doi: 10.1007/s00198-021-05900-y. Epub 2022 Apr 28. PMID 35478046
- [Result] Gullberg B, Johnell O, Kanis JA. World-wide projections for hip fracture. Osteoporos Int. 1997;7(5):407-13. doi: 10.1007/pl00004148. PMID 9425497
- [Result] Cooper C, Campion G, Melton LJ 3rd. Hip fractures in the elderly: a world-wide projection. Osteoporos Int. 1992 Nov;2(6):285-9. doi: 10.1007/BF01623184. PMID 1421796
- See also: National Institute of Arthritis and Musculoskeletal and Skin Diseases. (2022.12) Osteoporosis. National Institutes of Health(NIH). — https://www.niams.nih.gov/health-topics/osteoporosis
- See also: 中華民國骨質疏鬆症學會(2025 年 10 月 30 日)。2025 台灣成人骨質疏鬆防治之共識及指引。 — https://www.toa1997.org.tw/upload/news/224/171.pdf?v=251030161815